CLINICAL TRIAL: NCT06854198
Title: Novel Telehealth Technologies to Detect and Manage Glaucoma and Vision-threatening Eye Diseases in High-risk Populations
Brief Title: Glaucoma Screening to Enhance At-Risk Californians' Health
Acronym: G-SEARCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 24-43132; U01DP006820 (NIH)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma
Keywords: optical coherence tomography; tonometry; glaucoma; screening
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence; Manometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Screening (Experimental)
  Interventions: Other: Glaucoma screening with optical coherence tomography (OCT), color fundus photography, and tonometry
- Education (Active Comparator)
  Interventions: Other: Educational Brochure
- Delayed Education (No Intervention): The same as the Educational Brochure arm, but delivered at the conclusion of the study.

INTERVENTIONS:
Other: Glaucoma screening with optical coherence tomography (OCT), color fundus photography, and tonometry — Participants will be called and offered a screening appointment. At the appointment, visual acuity, OCT, color fundus photography, tonometry, and visual field testing will be performed. The images will be assessed for abnormalities. Participants meeting referral criteria will be referred for a comprehensive eye examination with an eye care provider.
  Arms: Screening
Other: Educational Brochure — A brochure about glaucoma screening will be mailed to participants. The brochure will include contact information of a staff member who can schedule an appointment for a comprehensive eye examination.
  Arms: Education

SUMMARY:
The vast majority of glaucoma cases in the United States go undetected and untreated until the late stages of the disease. Open-angle glaucoma is a progressive condition that is asymptomatic in its early to moderate stages and may be amenable to screening through telemedicine-based approaches. This study is a randomized trial to evaluate whether glaucoma screening with established tests (e.g., optical coherence tomography, fundus photography, and tonometry) is more effective for detecting undiagnosed glaucoma cases compared to education alone or delayed intervention.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the effectiveness of a telemedicine-based glaucoma screening program for detecting glaucoma. The investigators hypothesize that a mobile screening intervention incorporating optical coherence tomography (OCT), fundus photography, and tonometry will result in a greater number of new glaucoma diagnoses compared to education alone or delayed treatment.

Specific Aim 2: To determine whether a telemedicine-based glaucoma screening program provides benefits beyond glaucoma detection. The investigators hypothesize that (A) individuals randomized to the screening intervention will have higher rates of cataract surgery and distance vision correction one year after screening, and (B) those in the screening intervention will report higher vision-related quality of life one year after screening.

ELIGIBILITY:
Inclusion Criteria:

* Black people aged 50 years or older
* Hispanic people aged 65 years or older
* People with diabetes aged 50 years or older
* Must have been seen at the Federally Qualified Health Center (FQHC) within the past month

Exclusion Criteria:

* Patients without a valid phone number or mailing address
* Patients who have had an optometry appointment within the past year

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Glaucoma Diagnosis or Glaucoma Suspect Requiring Treatment | 3 months from randomization

SECONDARY OUTCOMES:
Cataract surgery | 12 months
  Self-reported cataract surgery
Eyeglasses | 12 months
  Self-reported purchase of new distance eyeglasses
Quality of Life survey | 12 months
  Self-reported quality of life on VisQol instrument

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Keenan, MD, MPH, Principal Investigator — University of California, San Francisco; Yvonne Ou, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
treatment arm, age, gender, results of diagnostic tests, 3-month and 12-month questionnaires
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the primary papers.
Access Criteria: Researchers interested in accessing imaging data from this project will submit requests to the investigators following instructions available at the repository. The study's co-PIs will approve requests with clear research questions and processes in place to ensure secure storage of images.